CLINICAL TRIAL: NCT01206530
Title: A Phase I/II Pharmacodynamic Study of Hydroxychloroquine in Combination With FOLFOX Plus Bevacizumab to Inhibit Autophagy in Colorectal Cancer
Brief Title: FOLFOX/Bevacizumab/Hydroxychloroquine (HCQ) in Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: UPCC 07210
Record Dates: First submitted 2010-09-16; First posted 2010-09-22 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Rectal Cancer; Colon Cancer; Metastasis; Adenocarcinoma
Keywords: histologically documented; advanced; metastatic; adenocarcinoma; colon; rectum
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms; Neoplasm Metastasis; Adenocarcinoma | interventions — Hydroxychloroquine; Oxaliplatin; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Hydroxychloroquine — Dose:600 or 800 mg Route:PO daily Treatment Administration: Daily
Drug: Oxaliplatin — Dose: 85mg/m2 Route: IV infusion over 2 hours Treatment Administration: Day 1
Drug: Leucovorin — Dose: 400mg/m2 Route IV infusion over 2 hours Treatment Administration: Day 1
Drug: 5-fluorouracil — Dose: 400mg/m2 Route: IV bolus immediately following leucovorin Treatment Administration Day 1
Drug: 5-fluorouracil — Dose: 2,400mg/m2 Route: IV continuous infusion over 46 hours immediately following bolus injection.
  Treatment Administration: Days 1-2
Drug: Bevacizumab

SUMMARY:
In this Phase I/II clinical trial, the investigators seek to pilot the addition of hydroxychloroquine (HCQ) to the standard front-line therapy of colorectal cancer, FOLFOX/bevacizumab. In toxicity terms, the investigators previous studies lead them to believe that a full dose (800mg) of HCQ will be well-tolerated in this setting. By starting at 600 mg, the investigators will ensure that the full dose is approached with an eye to safety, and if needed, the investigators will use the lower dose. Both doses achieve autophagy inhibition in our current studies.

DETAILED DESCRIPTION:
In this Phase I/II clinical trial, we seek to pilot the addition of HCQ to the standard front-line therapy of colorectal cancer, FOLFOX/bevacizumab. In toxicity terms, our previous studies lead us to believe that full dose (800mg) of HCQ will be welltolerated in this setting. By starting at 600 mg, we will ensure that the full dose is approached with an eye to safety, and if needed, we will use the lower dose. Both doses achieve autophagy inhibition in our current studies: for this reason, we are comfortable in including accrual to both dose-levels to the Phase II endpoints. If results are particularly striking, we will consider amending the study to expand accrual if the budget permits, but 25 patients permits an adequate assessment of activity of a novel regimen. The correlative endpoints of this trial are directed to the pharmacokinetics of HCQ, and pharmacodynamics of autophagy inhibition. We are currently constructing a population pharmacokinetic model of HCQ based on data from several ongoing trials, and the data from these patients will contribute to refining the model. We will analyze both measured and modelpredicted indices for their relationship to autophagy induction. Autophagy will be assessed as the accumulation of autophagocytic vesicles in the PMNs of treated patients, together with the induction of the expression of autophagyrelated proteins on western analysis, quantitated by densitometry. An exploratory correlative endpoint is the induction of metabolic changes as measured by 18FDG-PET. Our mechanistic hypothesis in this work is that the addition of HCQ will lead to a greater amount of cell death in the hypoxic regions of the tumor, that have increased as a consequence of bevacizumab treatment. We will document the rates of metabolic response as a consequence of treatment, as a therapeutic marker that may be related to the degree of autophagy inhibition. Finally, since we have demonistrated the key role of JNK1 in the induction of autophagy, we will analyze archival tumor materials to determine variability in this marker, as a baseline for potential future trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented advanced or metastatic adenocarcinoma of the colon or rectum.
* Patients must have measurable disease as defined by the RECIST criteria as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as 20 mm with conventionaltechniques on either CT of MRI. Marker (CEA) elevation alone is insufficient for entry.
* Patients may have had prior adjuvant treatment of advanced colorectal cancer. The prior treatment regimen must not have included bevacizumab but may have included oxaliplatin and the last dose of chemotherapy must have been 6 months prior to study entry. Patients with prior radiotherapy are acceptable. It must be at least 2 weeks since administration of radiation therapy and all signs of toxicty must have abated.
* Patients must be 18 years or older.
* Patients must have an ECOG performance status of 0-1.
* The following required Initial Laboratory Values should be obtained within 4 weeks of the start of treatment: Granulocytes 1,500/ml, Platelet Count 100,000/ml, Creatinine 1.5 x upper limit of normal, Bilirubin 1.5 x upper limit of normal, AST 5 x upper limit of normal Urine Urine protein:creatinine ratio 1.0 at screening
* Patients must not be pregnant or lactating as chemotherapy is thought to present substantial risk to the fetus/infant.
* Patients must have a life expectancy of greater than three months.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Major sugical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study. Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0.
* Patients with serious nonhealing wounds, ulcers, or bone fractures.
* Patients with a history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to Day 0
* Patients with a history of myocardial infarction, unstable angina, or cerebrovascular accident 6 months prior to registration.
* Patients with clinically significant peripheral vascular disease.
* Patients with New York Heart Association Class II or greater congestive heart failure (class II is defined as symptoms of fatigue, dyspnea or other symptoms with ordinary physical activity).
* Patients using oral or parenteral anticoagulation are not excluded provided they are on a stable dose of anticoagulant.
* Patients with pre-existing hypertension should be on a stable antihypertensive regimen and have a blood pressure 150/100 mmHg at the time of enrollement.
* Patients must not have known brain metastases because the study drug has not been adequately tested in this setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Response Rate
  We will use response as the primary efficacy marker to investigate the relationship between changes in autophagy markers and SUVs and the efficacy of treatment.

SECONDARY OUTCOMES:
Progression-free survival
  To evaluate the effects of baseline markers and treatment group on time to progression and survival, we will estimate propportional-hazards regression models. Time-to-event outcomes will be summarized with Kaplan-Meier survival curves.
Overall survival
  To evaluate the effects of baseline markers and treatment group on time to progression and survival, we will estimate propportional-hazards regression models. Time-to-event outcomes will be summarized with Kaplan-Meier survival curves.
Incidence of toxicity
  To evaluate the effects of baseline markers and treatment group on time to progression and survival, we will estimate propportional-hazards regression models. Time-to-event outcomes will be summarized with Kaplan-Meier survival curves.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. O'Dwyer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Mendonca Gorgulho C, Krishnamurthy A, Lanzi A, Galon J, Housseau F, Kaneno R, Lotze MT. Gutting it Out: Developing Effective Immunotherapies for Patients With Colorectal Cancer. J Immunother. 2021 Feb-Mar 01;44(2):49-62. doi: 10.1097/CJI.0000000000000357. PMID 33416261